CLINICAL TRIAL: NCT03647007
Title: Evidence of the Short- and Long-term Effects of a Residential Stay in a Danish Christmas Seal Home - With and Without a High-intensity Activity/Health Education (FIFA 11 for Health) Programme.
Brief Title: Short- and Long-term Health Effects of a Residential Stay in a Danish Christmas Seal Home.
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Peter Krustrup, Professor, University of Southern Denmark
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: Christmas Seal Home Project
Record Dates: First submitted 2018-08-20; First posted 2018-08-27 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Overweight
Keywords: fat percentage; physical fitness; well-being; small-sided games
MeSH Terms: conditions — Overweight | interventions — Health

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard group (No Intervention): The Standard programme on the Christmas Seal Homes.
- FIFA Group (Experimental): The Standard programme including FIFA 11 for Health programme - health knowledge on the football pitch.
  Interventions: Other: FIFA 11 for health

INTERVENTIONS:
Other: FIFA 11 for health — The training consists of various football exercises, such as passing, shooting, dribbling, etc., and small-sided games. The small-sided games are performed as e.g. 3v3 with small goals (2x5 m).
  Arms: FIFA Group

SUMMARY:
The purpose of the study is: (1) to evaluate the short-term effects of a 10-week residential stay in a Danish Christmas Seal Home on health, physical fitness, physical activity level, learning, sleep and well-being; (2) to investigate the long-term effects 3 and 12 months after the stay; and (3) to examine whether a special effort involving a high-intensity activity/health education programme (FIFA 11 for Health) increases the effects on physical fitness and health knowledge, learning capabilities, sleep patterns, well-being and adherence to a physically active lifestyle compared to the standard programme.

DETAILED DESCRIPTION:
Design Approx. 600 boys and girls aged 7-14 years are recruited from two Danish Cristmas Seal Homes (DCSHs) during 2018-2020. The design is a cross-over design at DCSH level over a two-year period with two intervention groups: a standard group (with the standard programme (SG)) and a standard + FIFA group (SG+). In SG+, the children, in addition to the standard programme, play recreational football for 2x45 min a week. In SG, the children perform the activities according to the regular schedule. In SG+, consist of different football exercises (dribbling, ball control, passing, etc.) and small-sided games with high intensity (3v3 to 5v5) using two goals. Every week, a specific football skill is linked to a health message, e.g. the skill of passing the ball to one another is linked to mutual respect and avoiding bullying.

Training protocol Recreational football The risk of injury for young players is markedly higher (5 times higher) in football match-play than in football training. While it is noted that muscle strains and twisting injuries in joints can also occur during training with small goals, the injury frequency for 10-year-old children in football training is approx. 5 per 1,000 training sessions, and hence low. Furthermore, the FIFA 11 for Health pilot study, which involved Danish 10-11-year-old schoolchildren, did not record any injuries during the training.

Tests and measurements The participants are tested at the start and end of their 10-week residential stay at the DCSH. Furthermore, there are follow-up tests 3 and 12 months after their stay. The four test days include measurements of physical fitness, physical performance, cognitive functions and questionnaires about health knowledge, well-being and sleep patterns. For further descriptions, see below.

Each test day, lasting approx. 4-5 hours, is planned in collaboration with DCSH staff and implemented by a member of the scientific group (human physiologists).

Anthropometric measurements: Body weight and standing and sitting height are measured using a portable body composition analyser (InBody 720) and an altimeter, respectively. The InBody 720 also provides an estimate of muscle mass and fat percentage. After a minimum of 10 min of resting in the supine position in a quiet room, measurements of resting heart rate and blood pressure are performed.

Balance and muscle strength/horizontal jumping performance: Balance performance is measured using the Stork test. It is measured on both legs, with the best of three attempts counting as the result. The child stands on the floor barefoot or in socks, eyes open with their weight on the entire sole of the supporting foot, arms on hips and the non-weight-bearing foot placed on the inside of the opposite knee. When the child has got their balance, the heel of the supporting foot is lifted and the time starts. The time stops for the following reasons:

* Hands/arms leave the hips.
* Supporting foot moves.
* Heel touches the floor.
* Foot resting on the knee is removed from the knee.

Explosive leg strength: Measured by a standing longitudinal jump. The starting position is with hands on hips and bent knees. The participants start the jump from behind a line on the floor with a two-footed take-off and land on their feet on a thin mat. The distance from the take-off to the point where the rear heel contacts the mat is noted and the best of two attempts counts. Standing longitudinal jumping is correlated with both upper- and lower-body strength tests in children and adolescents, and can therefore be considered as a general index for muscular fitness.

Aerobic fitness and intermittent performance: The original Andersen interval running test is used for indirect estimation of maximal oxygen uptake. The participants run back and forth between cones in a 20-m lane, touching the line between the cones at each end. After 15 s, the participant stops as quickly as possible (about two steps) and rests for 15 s. This procedure is followed for a total of 10 min. The 15-s periods are indicated by music, which stops during rest periods. All participants start and finish the test at the same time. The distance covered is recorded as the test result. This test has previously been performed in 6-13-year-olds, and no risks or adverse effects have been observed. The test is also validated for children in the age group 6-13 years.

Cognitive functions: During the four test rounds, the participants are tested using a computer-based objective cognitive test battery that has been validated and verified in the age group 10-18 years for measuring children's cognitive functions. The battery consists of four tests measuring reaction time, attention, visual learning and long-term memory, work memory and executive functions.

Metabolic markers: Saliva collected using a Salivette tube is used to indicate the level of hormone insulin. The insulin level may indicate an increased risk of insulin resistance and type 2 diabetes. Saliva samples are kept as cold as possible until they can be centrifuged. Samples are centrifuged and the supernatant stripped into cryo tubes and stored at -20 degrees, then -80 degrees.

Hair samples are taken for determination of long-term exposure to the biomarker cortisol. These consist of approx. 100 hairs cut as close to the scalp as possible. They are kept in an envelope until analysis.

Health knowledge and general and sports psychology measurements Questionnaires are used at baseline, at the end of the DCSH stay, and 3 and 12 months after the stay to examine the participants' health, well-being/mental health, ego and task orientation, cohesion, stress levels and sleep habits. During completion of the questionnaires, a supervisor is present to assist with any problems with reading and understanding. The participant's health knowledge is measured using a questionnaire that examines their learning and understanding of the 11 health messages. There is a total of 38 questions. The purpose of the questionnaire is to investigate how much the participant has learned about each of the 11 health messages in the programme.

The participant's well-being/mental health is measured using a PedsQL questionnaire as well as a Kids Screen questionnaire. The questionnaires, comprising 22 and 25 questions, respectively, aim to measure the well-being of the participant and cover a wide range of dimensions in well-being. A previous survey has tested the validity of the questions.

The participant's ego and task orientation is measured using the Task and Ego Orientation in Sport Questionnaire (TEOSQ). The questionnaire comprises 13 questions (7 for task and 6 for ego orientation) that are answered on a Likert scale of 1 to 5, where 1 is "strongly disagree" and 5 is "strongly agree". Task-oriented participants emphasise doing their best, experiencing progress and/or improving their skills, while ego-oriented participants measure themselves against others and emphasise being successful and better than others. The questionnaire has been validated and translated into Danish. TEOSQ has been used in Danish studies.

The participant's cohesion is measured using the Youth Sport Environment Questionnaire (YSEQ). The questionnaire comprises 12 questions that are answered on a Likert scale of 1 to 5, where 1 is "does not fit" and 5 is "fits completely". Cohesion describes how the participant perceives the class's solidarity regarding social aspects and its ability to solve tasks in unity. The questionnaire has been validated in English and the Danish version has been used in similar studies.

The Children's Sleep Habits Questionnaire (CSHQ) is used to assess the participant's sleep habits. The questionnaire is available in several versions comprising 33 or 26 questions for completion by the parents and the child, respectively. The questions are answered "usually" (5 to 7 times a week), "sometimes" (2 to 4 times a week) or "rarely" (0 to 1 time a week). The questionnaires clarify sleep habits, sleep disorders and consequences of disturbed sleep. The questionnaires have been validated in English, and the parents' version has been used in studies in Danish. The children's version will be used at baseline, at the end of the 10-week DCSH residential stay, and both 3 and 12 months after the stay, while the parents' version will be used at baseline and 3 and 12 months after the stay. The children's version is in English. Before the start of the study, the version will undergo a process of translation into Danish, back-translation into English and pre-testing with 5-10 children, and can thus be used as a self-reporting version.

The participant's stress levels are measured using the Strengths and Difficulties Questionnaire (SDQ). The self-completion version for the children has been validated in English. The questionnaire comprises 30 questions answered with "fails", "fits partially" or "fits well" within the last 6 months (baseline - afterwards, within the last month). The children's version will be used at baseline, after the DCSH stay, as well as both 3 and 12 months after the stay. The questionnaire reveals symptoms of emotional, behavioural, hyperactivity/concentration and social challenges. The parents' version has previously been used in studies with Danish youth (5-12 years). The parents' version will be used at baseline and 3 and 12 months after the stay.

Other measurements

In addition to the above test days, the following measurements are performed:

Continuous intensity measurements during training

Activity recordings are carried out frequently during the training intervention. Measurements are performed up to four times for approx. 50 participants from each DCSH, including pulse rate measurements (Polar Team 2), GPS measurements and accelerometer measurements to determine intensity and motion pattern analysis. At the training sessions where activity recordings are carried out, short questionnaires are also provided to measure perceived exertion and flow in relation to the training. In relation to accelerometer measurements, participants' daily activity level and sleep patterns are also recorded for up to 25% of participants during the intervention period.

Additional information Socioeconomic data, ethnicity and background details and health data are obtained via a parent-completed questionnaire. Absence lists, as well as results from school-related tests, are also obtained through the DCSH to exploit the large number of participants in various subgroup analyses.

ELIGIBILITY:
Inclusion Criteria:

* • Boys and girls aged 7-14 years undergoing a 10-week DCSH residential stay.

  * Informed consent from parents/legal guardian.
  * Willingness to participate in training and testing.

Exclusion Criteria:

* • Participants found by the researchers to be unsuited to following the procedures of the protocol and the training and testing programme.

Ages: 7 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 600 (Estimated)
Dates: Start 2018-09-11 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
changes in overweight | baseline, 10 weeks, follow-up - 3 and 12 months
  measurements of fat percentage, portable body composition analyser (InBody 720)

SECONDARY OUTCOMES:
aerobic fitness, measured with Andersen running test | baseline, 10 weeks, follow-up - 3 and 12 months
  The original Andersen interval running test is used for indirect estimation of maximal oxygen uptake.
health knowledge, questionnaires | baseline, 10 weeks, follow-up - 3 and 12 months
  The participant's health knowledge is measured using a questionnaire that examines their learning and understanding of the 11 health messages.
well-being, questionnaires | baseline, 10 weeks, follow-up - 3 and 12 months
  a PedsQL questionnaire as well as a Kids Screen questionnaire
BMI z-scores | baseline, 10 weeks, follow-up - 3 and 12 months
  weight (in kg) and height (in meters) will be combined to report BMI in kg/m^2

OTHER OUTCOMES:
muscle mass, portable body composition analyser (InBody 720) | baseline, 10 weeks, follow-up - 3 and 12 months
  The InBody 720 also provides an estimate of muscle mass and fat percentage.
sleep patterns, questionnaires | baseline, 10 weeks, follow-up - 12 months
  The Children's Sleep Habits Questionnaire (CSHQ)
daily activity patterns, accelerometre | baseline, 10 weeks, follow-up - 12 months
  accelerometre
insulin level | baseline, 10 weeks, follow-up - 12 months
  saliva samples
cortisol level | baseline, 10 weeks, follow-up - 12 months
  hair samples

CONTACTS AND LOCATIONS:
Overall Officials: Peter Krustrup, Principal Investigator — University of Southern Denmark
Locations (2):
- Denmark (2):
  - Skælskør Julemærkehjem, Skælskør, Region Sjælland
  - Kildemose Julemærkehjem, Ølsted, Region Sjælland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Pfeffer K, Nejst Larsen M, Cimenti C, Krustrup P, Ntoumanis N. Using the behaviour change intervention ontology to examine the inclusion, delivery and experience of behaviour change techniques in a youth health promotion programme. J Health Psychol. 2026 Jan 30:13591053251408386. doi: 10.1177/13591053251408386. Online ahead of print. PMID 41615742
- [Derived] Pfeffer K, Larsen MN, Heidler J, Moller TK, Tarantino G, Ntoumanis N, Krustrup P. The Long-Term Effects of a Combined Physical Activity and Health Education Programme on Well-Being for Socially Vulnerable Children and Adolescents. Scand J Med Sci Sports. 2025 Nov;35(11):e70171. doi: 10.1111/sms.70171. PMID 41263246

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-12-16): https://cdn.clinicaltrials.gov/large-docs/07/NCT03647007/Prot_SAP_002.pdf